CLINICAL TRIAL: NCT02245945
Title: Phase I Safety and Acceptability of Tenofovir 1% Gel in Adolescent Females
Brief Title: Safety and Acceptability of Tenofovir 1% Gel in Adolescent Females
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A14-130
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: HIV Prevention
Keywords: HIV; prevention
MeSH Terms: interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TFV 1% gel (Experimental): Participants will be instructed to use TFV 1% vaginal gel according to the BAT 24 regimen (2 gel doses) at least twice per week, regardless of sexual frequency.
  The BAT24 dosing regimen when used with sex is defined as one dose of gel within 12 hours before sex and a second dose of gel as soon as possible within 12 hours after sex and no more than two doses in a 24 hour period. Participants who do engage in sexual intercourse should use the BAT24 regimen with each sex act.
  If used without sex, the BAT24 dosing regimen is defined as 2 doses of gel administered 2-24 hours apart, with no more than two doses in a 24 hour period.
  Interventions: Drug: TFV 1% vaginal gel
- hydroxyethylcellulose (HEC) placebo gel (Placebo Comparator): Participants will be instructed to use HEC placebo gel according to the BAT 24 regimen (2 gel doses) at least twice per week, regardless of sexual frequency.
  The BAT24 dosing regimen when used with sex is defined as one dose of gel within 12 hours before sex and a second dose of gel as soon as possible within 12 hours after sex and no more than two doses in a 24 hour period. Participants who do engage in sexual intercourse should use the BAT24 regimen with each sex act.
  If used without sex, the BAT24 dosing regimen is defined as 2 doses of gel administered 2-24 hours apart, with no more than two doses in a 24 hour period.
  Interventions: Drug: HEC Placebo Gel

INTERVENTIONS:
Drug: TFV 1% vaginal gel — Tenofovir 1% gel is supplied as a clear, transparent, viscous gel packaged in pre-filled single use applicators. Each applicator contains 4.0 mL of tenofovir gel (equal to 4.4 gm) at a concentration of 1% (weight for weight) formulated in purified water with edetate disodium, citric acid, glycerin, methylparaben, propylparaben and hydroxyethylcellulose, and is pH adjusted to 4-5.
  Arms: TFV 1% gel
Drug: HEC Placebo Gel — Placebo gel contains hydroxyethylcellulose (HEC) as the gel thickener, purified water, sodium chloride, sorbic acid and sodium hydroxide. The gel is isotonic and formulated at a pH of 4.4. Each pre-filled applicator will contain approximately 4 mL of placebo gel for delivery.
  Arms: hydroxyethylcellulose (HEC) placebo gel

SUMMARY:
The purpose of this trial is to assess the safety and acceptability of Tenofovir (TFV) 1% gel in adolescent females over 12 weeks of a minimum of twice weekly dosing following the BAT24 regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 through 17 years, inclusive, as per site policy
* General good health (by volunteer history and per investigator discretion) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes)
* Able to communicate in spoken and written English
* Willing to following instructions regarding vaginal activity and vaginal products as follows:

  1. Willing to abstain from all vaginal activity, including intercourse, for 48 hours prior to Visit 2 and 48 hours prior to Visit 7
  2. Willing to abstain from the use of vaginal products other than the study product including spermicides, lubricants, and douches for the duration of study participation.

Note: Tampons may be used for menses, but pads should be used for any other intermenstrual spotting or bleeding.

* Assessment of onset and progression of puberty as measured by Tanner Stage 4 or 5
* History of consensual penile-vaginal intercourse (at least one episode in participant's lifetime)
* Negative urine pregnancy test
* Use of an effective method of contraception for at least the past 30 days (per participant report) and intended use for the duration of study participation. Effective methods include:

  1. Hormonal methods (excluding contraceptive ring)
  2. Intrauterine contraception (IUC)

Note: An IUC must be in place for at least 15 days prior to enrollment

* Willing to give voluntary assent, and comply with study procedures as required by the protocol assent and willing for parent/guardian to provide written informed consent for participation as per Institutional Review Board (IRB) requirements. Emancipated minors may give their own informed consent.

Exclusion Criteria:

* Known adverse reaction to study products (ever) or latex, per participant report
* Non-therapeutic injection drug use in the last 12 calendar months
* Post-exposure prophylaxis (PEP) for HIV-1 exposure within the last 6 calendar months
* Currently pregnant or within 30 days from the last pregnancy outcome.

Note: If recently pregnant must have had at least two spontaneous menses since pregnancy outcome.

* History of gynecological procedures (including genital piercing) on the external genitalia, vagina or cervix within the last 14 days
* Intention to become pregnant in the next 6 months
* Currently breastfeeding or having breastfed an infant in the last two months, or planning to breastfeed during the course of the study
* Positive for HIV
* Grade 2 or higher as per the Division of AIDS (DAIDS) Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009) of the following:

  1. Alanine transaminase (ALT), aspartate aminotransferase (AST)
  2. Creatinine
  3. Hemoglobin
  4. Platelet count
  5. Hepatitis B surface antigen (HBsAg)

Note: Otherwise eligible participants with an exclusionary test result(s) listed above may be re-tested a maximum of one time and if a non-exclusionary result is documented within the 30 days of providing informed consent, they may be enrolled.

* Clinically apparent Grade 2 or higher pelvic examination finding (observed by study staff) per the Female Genital Grading Table for Use in Microbicide Studies (Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009)

Note: 1) Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the Principal Investigator/designee is considered expected non-menstrual bleeding and is not exclusionary. 2) Otherwise eligible participants with exclusionary pelvic examination findings may be enrolled /randomized if improvement of findings to a non-exclusionary grade or to resolution can be documented within 30 days of providing informed consent for Screening.

* Current pelvic inflammatory disease (PID) or sexually transmitted infection requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines (e.g., Trichomonas vaginalis, Neisseria gonorrhea (GC), Chlamydia trachomatis (CT), or active herpes outbreak)
* Symptomatic vulvovaginal candidiasis, symptomatic bacterial vaginosis (BV) or urinary tract infection (UTI)

Note: Otherwise eligible participants with symptomatic vulvovaginal candidiasis, BV or UTI prior to genital sampling at Visit 2 will be offered treatment and may be continue in the study after completing treatment and all symptoms and findings have resolved.

* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, antifungals, antivirals (e.g., acyclovir or valacyclovir) or antiretrovirals (e.g., Viread®, Atripla®, Emtriva®, Complera®, Stribild®).

Note: Participants should avoid non-steroidal anti-inflammatory drugs (NSAIDs) except for treatment of dysmenorrhea during menses. Participants may use Tylenol® on an as-needed but not daily basis during the study.

* Participation in any other investigational trial (device, drug, or vaginal trial) within the last 30 days or planned participation in any other investigational trial during the study
* Any other condition that, in the opinion of the Principal Investigator (PI) or designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in genitourinary adverse events (AEs) | 24 hours after single dose; 1, 2, 4, 8 and 12 weeks during/after repeat dosing
  Number of genitourinary adverse events (AEs)
Changes in soluble markers of inflammation in cervicovaginal fluid (CVF) | Baseline; 24 hours after single dose; 12 weeks after repeat dosing
  changes in soluble markers of inflammation in cervicovaginal fluid (CVF)
Changes in vaginal microflora as assessed by Gram stain and semi-quantitative vaginal culture | Baseline and 12 weeks after repeat dosing
  Changes in vaginal microflora as assessed by Gram stain and semi-quantitative vaginal culture

SECONDARY OUTCOMES:
Responses to key questions on acceptability questionnaire | 2, 8 and 12 weeks during/after repeat dosing
  Responses to key questions on acceptability questionnaire
TFV concentration in plasma | 2 and 24 hours after single dose
  TFV concentration in plasma
TFV concentration in CVF | 24 hours after single does; 2, 4, 8, and 12 weeks during/after repeat dosing
  TFV concentration in CVF
Anti-HIV and anti-herpes simplex virus (HSV)-2 activity in the CVF | Baseline; 24 hours after single-dose; 12 weeks after repeat dosing
  Anti-HIV and anti-HSV-2 activity in the CVF
Real time adherence via internet-based diary | 12 weeks
  Real time adherence via internet-based diary
Biologic markers of adherence via returned empty applicators | 2, 4, 8 and 12 weeks during/after repeat dosing
  Biologic markers of adherence via returned empty applicators

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, MD, Study Director — CONRAD
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of Utah, Salt Lake City, Utah